CLINICAL TRIAL: NCT00499850
Title: A Phase I,Open Label Study to Assess the Safety and Tolerability of ZD6474 in Combination With 5-Fluorouracil, Leucovorin and Oxaliplatin (mFOLFOX6) as First and Second Line Therapy in Patients With Advanced Colorectal Adenocarcinoma.
Brief Title: Phase I FOLFOX Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00037
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Advanced Colorectal Carcinoma
Keywords: ZD6474; FOLFOX; colorectal; adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — vandetanib; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: ZD6474 (vandetanib) — once daily oral dose
  Other Names: ZACTIMA™
Drug: 5-Fluorouracil — intravenous infusion
  Other Names: 5-FU
Drug: Leucovorin — intravenous infusion
Drug: Oxaliplatin — intravenous infusion

SUMMARY:
A Phase I,open label study to assess the safety and tolerability of ZD6474 in combination with 5-Fluorouracil, Leucovorin and Oxaliplatin (mFOLFOX6) as first and second line therapy in patients with advanced colorectal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed locally advanced, recurrent or metastatic colorectal adenocarcinoma (Stage IV)
2. WHO performance status 0-1
3. one or more measurable lesions min 10mm by spiral CT or min 20mm by conventional techniques

Exclusion Criteria:

1. Brain metastasis or spinal cord compression unless irradiated at least 4 weeks before entry and stable
2. last dose of prior chemotherapy discontinued at least 4 weeks before start study treatment
3. prior unanticipated severe reaction to oxaliplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-08; Primary Completion 2006-06 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ZD6474 in combination with 5-Fluorouracil, Leucovorin and Oxaliplatin | Assessed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- Australia (4):
  - Research Site, East Melbourne
  - Research Site, Footscray
  - Research Site, Heidelberg
  - Research Site, Parkville